CLINICAL TRIAL: NCT06114134
Title: The Effect of Fenobet® Capsules (Fenugreek Seed Extract) on Glycemic Status, Lipid Pattern and Anthropometric Indices in People With Metabolic Syndrome: a Randomized, Double-blind, Controlled Clinical Trial.
Brief Title: The Effects of Fenugreek Extract (Fenobet) on Metabolic Syndrome
Acronym: Fenobet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nazli Namazi, Assistant Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 97-1151
Record Dates: First submitted 2023-10-09; First posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Metabolic Syndrome; Complementary Therapies; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fenugreek extract (Experimental): Participants in this group will receive fenugreek extract capsules (500 mg/day, three times a day, 30 minutes before each main meal) along with common treatments
  Interventions: Dietary Supplement: Fenobet
- Placebo (Placebo Comparator): Participants in this group will receive starch with added color (similar to the color of fenugreek extract) capsules (with the same size and color of fenugreek) (500 mg/day, three times a day, 30 minutes before each main meal) along with common treatments
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fenobet — receiving fenugreek extract (3 capsules of 500 mg, 1 capsule half an hour before meals)
  Arms: Fenugreek extract
Dietary Supplement: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The current study is a three-blind, randomized clinical trial study that will be conducted on 60 people with metabolic syndrome. The eligible participants were allocated randomly to one of the two study groups (Fenobet, Placebo). Then, the eligible people were in one of two groups 1) receiving fenugreek extract, 2), receiving placebos and were examined for 8 weeks. At baseline and after two months of intervention, biochemical parameters, and anthropometric indices will be measured.

DETAILED DESCRIPTION:
The current study is a three-blind, randomized clinical trial study that will be conducted on 60 people with metabolic syndrome. According to the ATP criteria, a person who has at least 3 of the following 5 components was considered as metabolic syndrome.

After providing the necessary information about the study to patients, written informed consent will be obtained from eligible volunteers.

Inclusion criteria:

* People with metabolic syndrome
* Fasting sugar above 100 mg/dL
* Both men and women
* Age range 20-60 years Exclusion criteria
* Injection of insulin or liraglutide
* People under 20 years old and over 60 years old
* having chronic cardiovascular diseases, chronic liver and kidney diseases, uncontrolled thyroid disorders and malignancies including cancer
* Taking herbal medicines or herbs to control blood sugar and fat in the last 6 months
* Patients who are treated with a special diet such as vegetarianism or a special exercise program.
* Allergy
* Pregnant and lactating women The participants were allocated randomly to one of the two study groups (Fenobet, Placebo) by a random number table. Then, the eligible people were in one of two groups 1) receiving fenugreek extract (3 capsules of 500 mg, 1 capsule half an hour before meals), 2), receiving placebos (3 capsules of 500 mg, 1 capsule half an hour before meals) and were examined for 8 weeks. It is worth noting that the participants were asked not to change their physical activity and diet during the study and to report any changes in the type and dosage of the drug to the researchers. The capsule and container intended for the placebo will be exactly the same size and color as the fenugreek capsule and a dark container will be chosen for the capsules. At baseline and after two months of intervention, biochemical parameters (fasting blood sugar, HbA1C, lipid profile, C-reactive protein), and anthropometric indices (weight, body mass index, waist circumference, Hip circumference) will be measured.

ELIGIBILITY:
Inclusion Criteria:

People with metabolic syndrome

* Fasting sugar above 100 mg/dL
* Both men and women
* Age range 20-60 years

Exclusion Criteria:

* Injection of insulin or liraglutide
* People under 20 years old and over 60 years old
* having chronic cardiovascular diseases, chronic liver and kidney diseases, uncontrolled thyroid disorders and malignancies including cancer
* Taking herbal medicines or herbs to control blood sugar and fat in the last 6 months
* Patients who are treated with a special diet such as vegetarianism or a special exercise program.
* Allergy
* Pregnant and lactating women

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2023-12-15 (Estimated); Study Completion 2024-02-20 (Estimated)

PRIMARY OUTCOMES:
Fasting blood sugar (FBS) | baseline and 2 months
  Fasting blood sugar in mg/dL will be reported
Hemoglobin A1C (HbA1C) | baseline and 2 months
  HbA1C will be reported in percentage

SECONDARY OUTCOMES:
Lipid profile | baseline and 2 months
  Total Cholesterol
Lipid profile | baseline and 2 months
  Triglyceride
Lipid profile | baseline and 2 months
  High-density Cholesterol (HDL-C)
Lipid profile | baseline and 2 months
  Low-Density Cholesterol (LDL-C)
Antropometric Indices | baseline and 2 months
  Weight
Antropometric Indices | baseline and 2 months
  Body Mass Index
Antropometric Indices | baseline and 2 months
  Waist Circumference
Antropometric Indices | baseline and 2 months
  Hip Circumference

IPD SHARING:
Plan to Share IPD: No